CLINICAL TRIAL: NCT04140695
Title: A Randomized, Double-blind, Placebo-controlled, Efficacy Study of the Neurokinin-1 Receptor Antagonist VLY-686 in Patients With Atopic Dermatitis
Brief Title: Evaluating the Effects of Tradipitant vs. Placebo in Atopic Dermatitis (EPIONE2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-3102; EPIONE2 (Other: Vanda Pharmaceuticals Inc.)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: Chronic Pruritus; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): Oral Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — BID
  Arms: Tradipitant
Drug: Placebo — BID
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to be conducted in the United States in subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female patients aged 18 - 70 years (inclusive);
* Diagnosed with atopic dermatitis;
* Suffering from chronic pruritus;
* Body Mass Index (BMI) of ≥18 and ≤40 kg/m2

Exclusion Criteria:

* Chronic pruritus due to condition other than atopic dermatitis (AD);
* A positive test for drugs of abuse at the screening or evaluation visits;
* Exposure to any investigational medication in the past 60 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Vanda Investigational Site, Hoover, Alabama
  - Vanda Investigational Site, Tempe, Arizona
  - Vanda Investigational Site, Encino, California
  - Vanda Investigational Site, Fountain Valley, California
  - Vanda Investigational Site, Laguna Hills, California
  - Vanda Investigational Site, Lomita, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, Clearwater, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Tampa, Florida
  - Vanda Investigational Site, Savannah, Georgia
  - Vanda Investigational Site, Boise, Idaho
  - Vanda Investigational Site, Chicago, Illinois
  - Vanda Investigational Site, Normal, Illinois
  - Vanda Investigational Site, Skokie, Illinois
  - Vanda Investigational Site, Plainfield, Indiana
  - Vanda Investigational Site, Crowley, Louisiana
  - Vanda Investigational Site, Timonium, Maryland
  - Vanda Investigational Site, Fort Gratiot, Michigan
  - Vanda Investigational Site, Saint Joseph, Missouri
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Omaha, Nebraska
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Berlin, New Jersey
  - Vanda Investigational Site, Hoboken, New Jersey
  - Vanda Investigational Site, Verona, New Jersey
  - Vanda Investigational Site, Kew Gardens, New York
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, The Bronx, New York
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Oklahoma City, Oklahoma
  - Vanda Investigational Site, Tulsa, Oklahoma
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Johnston, Rhode Island
  - Vanda Investigational Site, Spartanburg, South Carolina
  - Vanda Investigational Site, Dallas, Texas
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Mesquite, Texas
  - Vanda Investigational Site, South Jordan, Utah
  - Vanda Investigational Site, South Burlington, Vermont
  - Vanda Investigational Site, Alexandria, Virginia
  - Vanda Investigational Site, Newport News, Virginia
  - Vanda Investigational Site, Norfolk, Virginia
  - Vanda Investigational Site, Spokane, Washington

REFERENCES:
- See also: Study Webpage — http://advandastudy.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 43 | 44
Completed | 33 | 32
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (14.63) | 39.2 (15.10) | 40.4 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 30 | 28 | 58
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 5 | 3 | 8
  Black or African American | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 22 | 28 | 50
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Worst Itch Numeric Rating Scale (WI-NRS) Responder Rate at Week 2
Description: The WI-NRS responder is defined as a patient achieving at least 4 points reduction from baseline in weekly average of diary WI-NRS. Responses were measured on a scale of 0 - 10, with 0 being "no itch" and 10 being the "worst itch imaginable".
Time Frame: 2 weeks
Population: All participants randomized (1:1) to placebo or tradipitant.
Measure: Count of Participants; unit: Participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 42 | 43
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent through study completion (approximately 14 weeks) regardless of seriousness or relationship to investigational product. Patients with non-serious AEs that are ongoing at the patient's last study visit must be followed until resolution or for 30 days after the patient's last study visit, whichever comes first.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/44
Other Adverse Events (participants affected / at risk) | 13/43 | 10/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tradipitant (N=43) | Placebo (N=44)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tradipitant (N=43) | Placebo (N=44)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Chlamydial Infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Angular Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feces Discolored (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Liver Function Test Increased (Investigations) | 0 (0) | 1 (1)
Periorbital Oedema (Eye disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was discontinued early and therefore the study was not powered for appropriate examination of primary and secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04140695/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT04140695/SAP_001.pdf